CLINICAL TRIAL: NCT03007056
Title: Effect of High-flow Nasal Cannula Therapy on Exposure to Nasal Continuous Positive Airway Pressure in Very Preterm Infants
Brief Title: High Flow Nasal Cannula in Preterm Infants
Acronym: HIFLO
Status: Completed | Type: Observational
Sponsor: Hôpital de la Croix-Rousse (Other)
Responsible Party: Principal Investigator, Jean-charles PICAUD, MD, PhD, Professor of pediatrics, Hôpital de la Croix-Rousse
Other Study IDs: HIFLO
Record Dates: First submitted 2016-11-01; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Prematurity; Extreme
Keywords: high flow nasal cannula; nasal continuous positive airway pressure; noninvasive ventilatory support; newborn developmental care; bronchopulmonary dysplasia; weaning; pain; length of stay
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Period 1: year 2011 nCPAP
- Period 2: year 2014 nCPAP and high flow nasal cannula
  Interventions: Other: High flow nasal cannula

INTERVENTIONS:
Other: High flow nasal cannula — High flow nasal cannula added to the therapeutic arsenal in neonatal care
  Other Names: HFNC
  Groups: Period 2

SUMMARY:
The HIFLO study evaluates the impact of HFNC oxygen therapy on duration of nCPAP therapy, oxygen therapy and hospitalization. The cost of use of CPAP and two HFNC devices are also evaluated.

DETAILED DESCRIPTION:
Nasal continuous positive airway pressure (nCPAP) is widely used in preterm infants as it is efficient, but it creates an unfavorable environment for preterm infants. Indeed is a primary source of continuous noise in neonatal units and causes discomfort, pain, skin lesions. High flow nasal cannula (HFNC) introduced more recently in neonatal care supplies high allowing for carbon dioxide nasopharyngeal wash-out, reduction of work of breathing and is well tolerated. HFNC could help to improve the environment of preterm infants by reducing deleterious stimuli (noise, pain, discomfort) and by facilitating the contact between parents and babies. Efficacy of HFNC seems to be similar to other non-invasive respiratory supports for preventing treatment failure, death and bronchopulmonary dysplasia. The benefits of HFNC implementation was only slightly analyzed in extremely preterm infants. the place of HFNC is becoming increasingly important in neonatology and could help to improve the quality of care. Few HFNC devices are available but their cost of use has not been evaluated in Europe.

HIFLO study aimed to assess the impact of HFNC therapy introduction, on exposure to nCPAP and on the duration of oxygen therapy and hospital stay in preterm infants and in a subgroup of extremely preterm infants. The investigators also aim to evaluate the cost of use of nCPAP and HFNC using two different devices.

ELIGIBILITY:
Inclusion Criteria:

* Infants born before 32 weeks of gestational age
* Birth weight below 1500 g
* Infants hospitalized within the first 48 hours of life
* Infants discharged home from our unit

Exclusion Criteria:

* Infants transferred to another unit
* Infants with a severe malformation
* Infants requiring surgery

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All preterm infants born during year 2011 and year 2014, before 32 weeks of gestational age (GA) or with a birth weight below 1500 g, hospitalized within the first 48 hours of life in the tertiary care unit at Croix-Rousse Hospital, Lyon, France and discharged home from the unit.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Duration of exposure to nCPAP, expressed in days in the population of very preterm infants. | 2 years
  The study aim to compare two periods, before and after HFNC implementation. During the first period, in 2011, nCPAP (Infant FlowSiPAP) was used as a first-line non-invasive respiratory support. During the second period, in 2014, the use of HFNC support was established as soon as it was possible instead of nCPAP for prevention of apnea, or after extubation, and sometimes in infants with moderate respiratory distress syndrome treated without surfactant. Demographic characteristics, antenatal data, birth characteristics and neonatal morbidities, non-invasive ventilation oxygen administration and HFNC, postnatal steroid therapy, total duration of hospital stay, will be collected from our electronic standardized patient record in which they are prospectively encoded. Simple and multiple linear regression analyses will be used to evaluate the difference of nCPAP therapy duration between Group 1 and Group 2 after adjustment on potential cofactors.

SECONDARY OUTCOMES:
Duration of oxygen therapy (expressed in days) in the population of very preterm infants. | 2 years
  The study aim to compare two periods, before and after HFNC implementation. During the first period, in 2011, nCPAP (Infant FlowSiPAP) was used as a first-line non-invasive respiratory support. During the second period, in 2014, the use of HFNC support was established as soon as it was possible instead of nCPAP for prevention of apnea, or after extubation, and sometimes in infants with moderate respiratory distress syndrome treated without surfactant. Demographic characteristics, antenatal data, birth characteristics and neonatal morbidities, non-invasive ventilation oxygen administration and HFNC, postnatal steroid therapy, total duration of hospital stay, will be collected from our electronic standardized patient record in which they are prospectively encoded. Simple and multiple linear regression analyses will be used to evaluate the difference of nCPAP therapy duration between Group 1 and Group 2 after adjustment on potential cofactors.
Duration of hospital stay (expressed in days) in the population of very preterm infants. | 2 years
  The study aim to compare two periods, before and after HFNC implementation. During the first period, in 2011, nCPAP (Infant FlowSiPAP) was used as a first-line non-invasive respiratory support. During the second period, in 2014, the use of HFNC support was established as soon as it was possible instead of nCPAP for prevention of apnea, or after extubation, and sometimes in infants with moderate respiratory distress syndrome treated without surfactant. Demographic characteristics, antenatal data, birth characteristics and neonatal morbidities, non-invasive ventilation oxygen administration and HFNC, postnatal steroid therapy, total duration of hospital stay, will be collected from our electronic standardized patient record in which they are prospectively encoded. Simple and multiple linear regression analyses will be used to evaluate the difference of nCPAP therapy duration between Group 1 and Group 2 after adjustment on potential cofactors.
Duration of exposure to nCPAP (expressed in days) in extremely preterm infants. | 2 years
  It will be the same evaluation than in whole population, but in extremely preterm infants borm before 29 weeks gestational age.
The cost of use (expressed in Euros) of nCPAP and HFNC using two different devices. | 2 years
  Cost analysis will be carried out for the three devices: Infant Flow SiPAP, OptiFlow and Precision Flow, including all consumables. To evaluate the costs these devices will be used as recommended by the manufacturers.The calculated costs will be based on an example of three devices in constant use on a 7-day cycle change of the circuits for the Opti-Flow device, and 30-day cycle change for Precision Flow device. Actual costs will be expressed as price per patient per week.

CONTACTS AND LOCATIONS:
Overall Officials: jean-charles picaud, MD, PhD, Principal Investigator — Hopital de la croix rousse
Locations (1):
- Hopital de la croix rousse, Lyon, France

IPD SHARING:
Plan to Share IPD: No